CLINICAL TRIAL: NCT04834310
Title: Postoperative Antibiotics Following Primary and Secondary Breast Augmentation: A Double-Blinded, Randomized Trial
Brief Title: Postoperative Antibiotics Following Primary and Secondary Breast Augmentation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Do not have adequate funding to proceed with project.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Karie Villanueva, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCLA PRS
Record Dates: First submitted 2021-04-03; First posted 2021-04-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Surgical Site Infection; Capsular Contracture Associated With Breast Implant; Antibiotic Resistant Infection; Antibiotic Side Effect
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Clindamycin; Cephalexin

STUDY DESIGN:
Intervention Model Description: The study will be designed as a non-inferiority trial with two parallel groups: the experimental group will receive an intraoperative dose of antibiotics followed by oral antibiotics for 5 days postoperatively (Cephalexin 500 mg QID or Clindamycin 300 mg QID, if Penicillin allergic) while the control group will receive an intraoperative dose of antibiotics (Cefazolin 1 g or 2 g, or Clindamycin 600 mg or 900 mg, if Penicillin allergic, higher doses provided if BMI > 30 kg/m2) followed by a placebo for 5 days postoperatively.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed prior to surgery, and an assigned coordinator will generate group assignments. Patients and surgeons will be blinded to the study before randomization takes place. However, surgeons will have access to information following medication dispensation in case any complications arise so that the provider can carry out appropriate interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intraoperative and Postoperative Antibiotics (Experimental): The experimental group will receive an intraoperative dose of antibiotics, which is standard protocol at our institution, followed by oral antibiotics for 5 days postoperatively.
  Interventions: Drug: Cefazolin; Drug: Cephalexin
- Intraoperative Antibiotics and Placebo (Placebo Comparator): The control group will receive an intraoperative dose of antibiotics, which is standard protocol at our institution, followed by a placebo for 5 days postoperatively
  Interventions: Drug: Cefazolin; Other: Placebo

INTERVENTIONS:
Drug: Cefazolin — All patients will receive an intraoperative dose of IV Cefazolin 2 g (re-dose after 4 hours) or IV Clindamycin 600mg (re-dose after 6 hours) for penicillin allergic patients.
  Other Names: Ancef; Clindamycin; Cleocin
Drug: Cephalexin — The experimental group will receive a postoperative 5-day course of Cephalexin 500 mg QID or Clindamycin 300 mg QID for penicillin allergic patients. All capsules will be encapsulated with size 00 dark-colored capsules compounded by the UCLA Investigational Pharmacy.
  Other Names: Keflex; Clindamycin; Cleocin
  Arms: Intraoperative and Postoperative Antibiotics
Other: Placebo — The placebo group will receive a postoperative 5-day course of placebos (sugar capsules). All capsules will be encapsulated with size 00 dark-colored capsules compounded by the UCLA Investigational Pharmacy.
  Arms: Intraoperative Antibiotics and Placebo

SUMMARY:
Postoperative antibiotics are routinely used for implant-based breast augmentation at the investigators' institution. From 2017-2019, the investigators' institution has conducted approximately 270 primary and secondary breast augmentation procedures. Current plastic surgery literature does not provide recommendations for antibiotic prophylaxis following implant-based breast procedures. Despite controversy surrounding their utility during the postoperative course, postoperative antibiotics have become commonplace for many plastic surgeons. To date, strong scientific evidence supporting this practice is minimal and based largely on anecdotal evidence and limited studies, including poorly controlled retrospective and non-blinded prospective series. The goal of this study is to conduct a prospective randomized trial to assess whether extended antibiotic prophylaxis is necessary to prevent infection and long-term complications (e.g. capsular contracture) in patients undergoing augmentation mammoplasty with implants. The investigators' anticipate that extended antibiotic prophylaxis is not required. The rationale for discontinuing postoperative antibiotics is based on the following: (1) a single dose of preoperative intravenous antibiotics has been demonstrated to be sufficient prophylaxis for most breast surgeries and (2) there are patient safety concerns associated with prolonged antimicrobial use such as the development of resistant bacterial strains and clostridium-related infections. Concrete evidence that extended antibiotic prophylaxis is not required would encourage plastic surgeons to practice better antibiotic stewardship and help stymie the rise of drug-resistant organisms.

DETAILED DESCRIPTION:
The investigators will perform a randomized, double-blinded, placebo-controlled trial at University of California Los Angeles Ronald Reagan Medical Center for patients undergoing primary and secondary breast augmentation between 2021-2025. The study will be added to a research registry before patient enrollment begins (i.e. www.clinicaltrials.gov) with study methods and results presented in the manner recommended by the CONSORT statement (available at www.consort-statement.org). The study will be designed as a non-inferiority trial with two parallel groups: the experimental group will receive an intraoperative dose of antibiotics followed by oral antibiotics for 5 days postoperatively (Cephalexin 500 mg four times per day or Clindamycin 300 mg four times per day, if Penicillin allergic) while the control group will receive an intraoperative dose of antibiotics (Cefazolin 1 g or 2 g, or Clindamycin 600 mg or 900 mg, if Penicillin allergic, higher doses provided if BMI > 30 kg/m2) followed by a placebo for 5 days postoperatively. Inclusion criteria will include: females and transgender females 18 years or older, patients undergoing primary breast augmentation, breast augmentation-mastopexy, and secondary breast augmentation with subglandular or submuscular implants. Secondary breast augmentation will include patients undergoing implant exchange secondary to capsular contracture and implant rupture. Exclusion criteria will include refusal or inability to consent, patients with biopsy-proven breast cancer, patients undergoing expander-based and autologous flap breast reconstruction following mastectomies, history of chest radiation, and the presence of active infection at the time of surgery. Patients who fail to take the placebos or antibiotics provided in the study for any reason, miss postoperative visits, and/or withdraw consent at any stage of the study will also be excluded.

For the analysis, the investigators plan to obtain hospital records with intraoperative procedural and postoperative clinic notes. Demographic information including gender, body mass index, comorbidities, smoking use, and prior breast surgeries will be collected and used for analysis. Power analysis for statistical equivalency using 8% infection rate yields a required sample size of 164 total patients, with planned 82 patients per group (i.e. experimental and control). This would provide 80 percent power at a significance level of 5 percent. The experimental group will consist of patients who receive an intraoperative dose of antibiotics followed by oral antibiotics for 5 days postoperatively. The control group includes patients who receive an intraoperative dose of antibiotics followed by a placebo for 5 days postoperatively. All medications and placebos will be formulated, compounded and dispensed by the University of California Los Angeles Investigational Research Pharmacy. An appointed Data and Safety Monitoring Board (DSMB) will monitor data and safety as recommended by the Investigational Review Board (IRB).

Antibiotics of choice include intravenous Cefazolin and oral Cephalexin. Intravenous and oral Clindamycin will be made available for subjects who are allergic to Penicillin. Subject allocation will be based on a 1:1 ratio for each group. Surgeons, nursing, and administrative staff will be responsible for recruitment. Prior to surgery, patients will be given a consent form to explain their involvement in the randomized trial. The consent process will inform the participant about details of the study and indicate participation is voluntary. They will also be given the risks, benefits, alternatives, and confidentiality of their information with proceeding with the study. Risks discussed with participants will include those associated with antibiotic use, including gastrointestinal symptoms, yeast infections, allergic reactions, development of resistant bacterial strains, and clostridium-related infections. Potential risks associated with no antibiotic use (i.e. placebo group), include infection. The interventions to protect those affected by these risks include hospital admission as detailed in the informed consent under the section "Office of the Human Research Protection Program (OHRPP)," and the option to opt out of the study. There are no medical benefits with participating in the study. However, participants will be informed that the results may contribute to the body of knowledge around postoperative antibiotics, and improve surgical protocols and postoperative care.

Randomization will be performed prior to surgery, and an assigned study coordinator will generate group assignments. Patients and surgeons will be blinded to the study before randomization takes place. However, surgeons will have access to information following medication dispensation in case any complications arise so that the provider can carry out appropriate interventions. Review of the rate of subject accrual and compliance will occur monthly during the recruitment phase. An interim analysis will be performed on the primary endpoint when 50% of patients have been randomized and have complete their 6-month follow up period. An independent statistician blinded to treatment allocation will perform the analyses. The statistician will report to DSMB who will have unmasked access to all data. Interim analysis will be used to inform stopping guidelines and trial adaptations (e.g. sample size re-estimation, alteration to the proportion of participants allocated to each study group, and changes to eligibility criteria). The Principal Investigator (PI) will be responsible for ensuring participants' safety on a daily basis. The DSMB will act in an advisory capacity to monitor participant safety, evaluate the progress of the study, and review procedures for maintaining the confidentiality, quality, management, and analysis of the data.

An adverse event will be any untoward medical occurrence in a subject without regard to the possibility of a causal relationship. Adverse events will be collected after the subject has provided consent and enrolled in the study. All adverse events occurring after entry into the study and up to their first postoperative visit will be recorded. A serious adverse event for this study is any untoward medical occurrence that is believed by the investigators to be causally related to study-drug and results in any of the following: life-threatening condition (i.e. immediate risk of death); severe or permanent disability, prolonged hospitalization, or a significant hazard as determined by the DSMB. Investigators will determine relatedness of an event to study based on a temporal relationship, as well as whether the event is unexpected or unexplained given the subject's clinical course, previous medical conditions, and concomitant medications. All adverse and severe events related to antibiotic use, including anaphylaxis requiring hospital admission and/or resulting in death, will be monitored through patient examination and chart review. Furthermore, events that meet criteria for an adverse and serious adverse will be reported to the IRB.

Six plastic surgeons will be involved in the study and will utilize a standardized surgical protocol. Initial follow up visits will be arranged within 1-2 weeks following surgery. Data on adherence to the treatment protocol will be collected monthly by research staff and reviewed quarterly by the Principal Investigator and the study statistician. Adherence of participants will be evaluated by inquiring about completion of antibiotics or placebos at each postoperative visit. During follow-up visits, inquiry will be made to assure patients receive their antibiotics or placebos. This information along with any post-operative complications will be transferred onto the patient's electronic medical record accordingly. Primary outcomes including surgical site infection, secondary outcomes (e.g. hematoma, seroma, wound dehiscence, implant loss, and capsular contracture), and antibiotic-related complications (e.g. antibiotic resistance, diarrhea, clostridium infection, yeast infections, rash, urinary tract infections, and gastrointestinal upset) will be documented. Surgical site infections will be determined by the surgeon however will be defined by the presence of the following signs and symptoms: fevers, purulent drainage, pain, tenderness, localized edema, heat, erythema, positive wound cultures, and leukocytosis. Study endpoints will include diagnosis of surgical site infection, development of secondary outcomes, and subject death or loss to follow-up. Follow-up will be continued until all patients have reached one of the study endpoints. Statistical tests will be performed by a statistician using statistical software and determined after enough data has been generated to perform preliminary analysis. Threats to study validity include under recruitment of subjects, subjects lost to follow-up, subject non-compliance, and subject crossovers. This study will be stopped prior to its completion if: the intervention is associated with adverse effects that call into question the safety of the intervention; difficulty in study recruitment or retention will significantly impact the ability to evaluate the study endpoints; any new information becomes available during the trial that necessitates stopping the trial; or other situations occur that might warrant stopping the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 year or older
* Participants undergoing primary breast augmentation with subglandular or submuscular implants
* Participants undergoing breast augmentation-mastopexy with subglandular or submuscular implants
* Participants undergoing secondary breast augmentation with subglandular or submuscular implants (i.e. patients undergoing implant exchange secondary to capsular contracture and implant rupture)

Exclusion Criteria:

* Refusal or inability to obtain consent from participants
* Participants with biopsy-proven breast cancer
* Participants undergoing expander-based breast reconstruction
* Participants undergoing autologous flap breast reconstruction
* Participants with history of chest radiation
* Participants with active infection at the time of surgery
* Participants who fail to take the placebos or antibiotics provided in the study for any reason
* Participants who miss postoperative visits
* Participants who withdraw consent at any stage of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with surgical site infection | 365 days following surgery
  Surgical site infections will be determined by the surgeon however will be defined by the presence of the following signs and symptoms: fevers, purulent drainage, pain, tenderness, localized edema, heat, erythema, positive wound cultures, and leukocytosis.

SECONDARY OUTCOMES:
Number of participants with hematoma | 365 days following surgery
  Fluid collection consisting of blood secondary to procedure identified by clinical exam and/or ultrasound.
Number of participants with seroma | 365 days following surgery
  Fluid collection consisting of serous fluid secondary to procedure identified by clinical exam and/or ultrasound.
Number of participants with wound dehiscence | 365 days following surgery
  Any re-opening of surgical incision following procedure which was closed primarily.
Number of participants with implant loss | 365 days following surgery
  Extrusion of implant or condition resulting in implant removal secondary to procedure.
Number of participants with antibiotic-related complications | 365 days following surgery
  Diarrhea, clostridium infection, yeast infections, rash, urinary tract infections, and gastrointestinal upset
Number of participants with antibiotic resistance | 365 days following surgery
  Local wound infections and fluid collections will be cultured and sent for identification and susceptibility. Resistant strains will be documented and treated with alternative antibiotics.

OTHER OUTCOMES:
Patient compliance | 365 days following surgery
  Patients will be asked during the first postoperative visit if they had taken their placebos or antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Karie Villanueva, MD, Principal Investigator — University of California, Los Angeles; Jaco Festekjian, MD, Study Chair — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chopra K, Gowda AU, McNichols CHL, Brown EN, Slezak S, Rasko Y. Antimicrobial Prophylaxis Practice Patterns in Breast Augmentation: A National Survey of Current Practice. Ann Plast Surg. 2017 Jun;78(6):629-632. doi: 10.1097/SAP.0000000000000942. PMID 27922894
- [Background] Hardwicke JT, Bechar J, Skillman JM. Are systemic antibiotics indicated in aesthetic breast surgery? A systematic review of the literature. Plast Reconstr Surg. 2013 Jun;131(6):1395-1403. doi: 10.1097/PRS.0b013e31828bd752. PMID 23416440
- [Background] Keramidas E, Lymperopoulos NS, Rodopoulou S. Is antibiotic prophylaxis in breast augmentation necessary? A prospective study. Plast Surg (Oakv). 2016 Fall;24(3):195-198. doi: 10.4172/plastic-surgery.1000976. Epub 2016 Aug 19. PMID 28439510
- [Background] LeRoy J, Given KS. Wound infection in breast augmentation: the role of prophylactic perioperative antibiotics. Aesthetic Plast Surg. 1991 Fall;15(4):303-5. doi: 10.1007/BF02273877. PMID 1950803
- [Background] Mirzabeigi MN, Mericli AF, Ortlip T, Tuma GA, Copit SE, Fox JW 4th, Moore JH Jr. Evaluating the role of postoperative prophylactic antibiotics in primary and secondary breast augmentation: a retrospective review. Aesthet Surg J. 2012 Jan;32(1):61-8. doi: 10.1177/1090820X11430830. PMID 22231414
- [Background] Gylbert L, Asplund O, Berggren A, Jurell G, Ransjo U, Ostrup L. Preoperative antibiotics and capsular contracture in augmentation mammaplasty. Plast Reconstr Surg. 1990 Aug;86(2):260-7; discussion 268-9. PMID 2195567